CLINICAL TRIAL: NCT05641155
Title: An Early Feasibility, Prospective, Exploratory Study Evaluating the Performance of Focused Multipolar Stimulation and Sound Coding Enhancements in Adult Cochlear Implant Recipients (SASC).
Brief Title: A Feasibility Study Evaluating the Performance of Focused Multipolar Stimulation and Sound Coding in Adults.
Acronym: SASC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI5781
Record Dates: First submitted 2022-11-09; First posted 2022-12-07 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Hearing Impairment, Sensorineural
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Adult Cochlear implant (Experimental): Adult cochlear implant recipients receiving different combinations of alternative modes and, sound coding parameters
  Interventions: Device: Focused Multipolar Stimulation (FMS) strategy

INTERVENTIONS:
Device: Focused Multipolar Stimulation (FMS) strategy — Adult cochlear implant recipients receiving different combinations of alternative modes and, sound coding parameters.

SUMMARY:
The purpose of this early feasibility study is to explore several facets of hearing performance that may show improvements for alternative modes of stimulation compared to Monopolar (MP stimulation) in cochlear implant recipients. This study will iteratively evaluate different parameter sets that intend to maximize hearing performance benefits within technical requirements. This study is exploratory in nature and will achieve its objectives through ongoing review and adjustment of device parameters and fitting

DETAILED DESCRIPTION:
Alternative modes of stimulation will be investigated that may improve spectral resolution through reduced cochlear spread of excitation and in turn provide enhanced speech perception and real-world clinical benefits over MP stimulation. The purpose of this study is to balance the clinical improvements of alternative modes of stimulation with technical and usability requirements for power usage. By iteratively evaluating different sets of stimulation and sound coding parameters, this study will determine device settings and fitting techniques. Measures of speech recognition, listening effort, neural responses, electrode placement, battery life, and usability acceptance will be obtained to evaluate clinical benefits

ELIGIBILITY:
Inclusion Criteria:

1) Candidate for unilateral cochlear implantation according to bilateral sensorineural hearing loss criteria, who has decided to proceed with implantation through routine processes.

a) Bilateral sensorineural hearing loss criteria for clinics in the United States: i) Ear to be implanted:

1. Moderate to profound sensorineural hearing loss, defined as a pure-tone average (PTA) (250 - 1000 Hz) ≥ 40 dB HL and a PTA (2000 - 8000 Hz) ≥ 65 dB HL
2. Aided word score ≤ 40% ii) Contralateral ear:

(1) PTA (500, 1000, 2000, and 4000 Hz) > 30 dB HL (2) Aided word score ≤ 80% b) Bilateral sensorineural hearing loss criteria for clinics in Belgium: i) Both ears:

1. PTA (500, 1000, 2000, and 4000 Hz) ≥ 70 dB HL for average of 3 out of 4 frequencies
2. Unaided phoneme score ≤ 50% on CVC in quiet at 70 dB SPL in free field
3. ABR peak ≥ 75 dB nHL

2) 18 years of age or older.

3) Fluent in the language used for speech testing.

4) Willing to comply with all investigational requirements.

5) Willing and able to provide written informed consent

-

Exclusion Criteria:

1. Previous or existing cochlear-implant recipient.
2. Severe or greater sensorineural hearing loss in the ear to be implanted prior to five years of age.
3. Duration of severe to profound hearing loss > 20 years in the ear to be implanted.
4. Ossification or other cochlear anomaly that might prevent complete insertion of the electrode array.
5. Diagnosis of auditory neuropathy.
6. Deafness due to lesions of the acoustic nerve or central auditory pathway.
7. Pregnant at the time of surgery.
8. Additional handicaps that would prevent or restrict participation in the audiological evaluations.
9. Unrealistic expectations on the part of the subject regarding the possible benefits, risks, and limitations that are inherent to the surgical procedure and prosthetic device.
10. Unable or unwilling to comply with the requirements of the clinical investigation as determined by the Investigator.
11. Investigator site personnel directly affiliated with this study and/or their immediate families; immediate family is defined as a spouse, parent, child, or sibling.
12. Cochlear employees or employees of Contract Research Organisations or contractors engaged by Cochlear for the purposes of this investigation.
13. Currently participating, or participated within the last 30 days, in another interventional clinical investigation/trial involving an investigational drug or device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-06-02 (Actual); Primary Completion 2025-02-06 (Actual); Study Completion 2025-12-08 (Actual)

PRIMARY OUTCOMES:
Mean difference across maximum map stimulation (C) levels | 10 weeks
  Mean difference across maps using alternative modes and sound coding parameters for the highest and average comfortable loudness level (clinical unit) (C-level).
Mean difference across Spectral resolution (QSMD) | 10 weeks
  Mean difference across maps using alternative modes and sound coding parameters for spectral resolution (% correct) (QSMD - Quick spectral modulation detection)
Mean difference across phoneme discrimination (LIT- Language independent test) | 10 weeks
  Mean difference across maps using alternative modes and sound coding parameters for phoneme discrimination (% correct) (LIT - Language independent test)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (2):
  - Rocky Mountain Ear Center, Englewood, Colorado
  - Denver Research and Technology Lab, Lone Tree, Colorado
- Belgium (3):
  - Universitair Ziekenhuis Leuven, Leuven, Leuven
  - Cochlear Technology Centre Belgium, Mechelen, Mechelen
  - ENT Department, Sint-Augutinus Antwerp, Wilrijk, Wilrijk

IPD SHARING:
Plan to Share IPD: No